CLINICAL TRIAL: NCT04171661
Title: SASS 3: Self-Assembled Skin Substitute (SASS) for the Treatment of Epidermolysis Bullosa
Brief Title: Self-Assembled Skin Substitute for the Treatment of Epidermolysis Bullosa
Acronym: SASS
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: The Hospital for Sick Children (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LOEX 019
Record Dates: First submitted 2019-11-19; First posted 2019-11-21 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Epidermolysis Bullosa Dystrophica
Keywords: Dystrophic Epidermolysis Bullosa; Recessive Dystrophic Epidermolysis Bullosa; Tissue Engineering; Skin Substitute
MeSH Terms: conditions — Epidermolysis Bullosa Dystrophica

STUDY DESIGN:
Intervention Model Description: n-of-one
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SASS (Experimental): SASS applied on chronic skin wounds as skin graft
  Interventions: Biological: SASS

INTERVENTIONS:
Biological: SASS — SASS applied on chronic skin wounds as skin graft

SUMMARY:
Single patient study. Patient diagnosed with dystrophic epidermolysis bullosa presenting chronic open wounds that are not responding to dressings, topical preparations (antimicrobials, antibiotics) and systemic agents (anti-inflammatory antibacterials). The Self-Assembled Skin Substitutes will be used to cover wounds.

ELIGIBILITY:
This clinical trial was custom designed for one patient

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2019-12-24 (Actual); Study Completion 2026-12-18 (Estimated)

PRIMARY OUTCOMES:
Percent reduction in wound surface area | 2 weeks
  Clinical assessment

SECONDARY OUTCOMES:
Graft failure | 2 weeks
  Clinical assessment
Number of subsequent re-transplantation | 3 years
  Number
Time (in weeks) to 50% reduction in the surface area of the wounds; | 3 years
  Clinical assessment
Time (in weeks) to complete healing | 3 years
  Clinical assessment
Changes in pain scores | 3 years
  10 point visual analog scale where 0 is none and 10 the worst pain
Changes in itch scores where 0 is none and 10 the worst itch | 3 years
  10 point scale

CONTACTS AND LOCATIONS:
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No